CLINICAL TRIAL: NCT02392585
Title: Triple Tourniquet vs. Single Tourniquet to Reduce Haemorrhage During Myomectomy: a Prospective Randomised Controlled Trial
Brief Title: Single or Triple Uterine Tourniquet at Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ragıp Atakan Al (Other)
Responsible Party: Sponsor-Investigator, Ragıp Atakan Al, Assoc.Prof, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATAUNİ23
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Uterine Myoma
Keywords: Leiomyoma of uterus; Hemostasis, Surgical; Prevention of Surgical Blood Loss; mechanical uterine tourniquet
MeSH Terms: conditions — Myofibroma | interventions — Tourniquets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single tourniquet (Active Comparator)
  Interventions: Procedure: Single tourniquet
- Triple tourniquet (Active Comparator)
  Interventions: Procedure: Triple tourniquet

INTERVENTIONS:
Procedure: Single tourniquet — Single tourniquet is tourniquet applied uterine isthmus to occlude the uterine arteries. For this purpose, a small opening is made in the avascular place of the broad ligament on either side of the uterine isthmus superior to the uterine vessels. A pediatric Foley catheter is threaded through the two holes and tied tightly anteriorly around the cervix at the level of the internal os.
  Arms: Single tourniquet
Procedure: Triple tourniquet — Triple tourniquet consist of two tourniquet applied both infundibulopelvic ligaments and one uterine isthmus to occlude the left and right ovarian vessels and to occlude the uterine arteries. For this purpose, a small opening is made in the avascular place of the broad ligament on either side of the uterine isthmus superior to the uterine vessels. A pediatric Foley catheter is threaded through the two holes and tied tightly anteriorly around the cervix at the level of the internal os.
  Through the same openings in the broad ligament each side a Foley catheter looped around the infundibulopelvic ligament lateral to the fallopian tube and ovary.
  Arms: Triple tourniquet

SUMMARY:
The aim of study is to compare triple tourniquet vs. single tourniquet to reduce blood loss at open myomectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Three or more uterine myoma
2. At least one myoma ≥ 8 cm, if there is less than three myoma

Exclusion Criteria:

1. Pedunculated myoma,
2. broad ligament myoma

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss at the end of myomectomy | 15 minutes postoperatively
  Surgical blood loss will be estimated by sum of the volume of suction fluid and blood loss quantitated by gravimetric method.
  Suction fluid will be measured at the end of operation and volume of irrigation fluid will be subtracted from total suction volume.
  ◦Surgical drapes, sponges and towels will be weighted before and just after surgery. The blood loss will be estimated as differences in gram by weighing when 1ml blood supposed as 1.06 gr.

SECONDARY OUTCOMES:
The amount of transfusions | 7 Days
  Erythrocyte transfusions will be allowed when haemoglobin dropped below 8 g/dL.
A change in hemoglobin | At baseline and 48 hours after surgery
Volume in drains | 7 days
  Drain will be removed when discharge drops below 50 ml/day
Peri-operative complications | 6 weeks
  Including but not limited to fever, pelvic infections, wound infections.
Total operation time | 5 minutes post operatively
  Skin to skin operation time
Tourniquet time | 5 minutes after tourniquet removed

OTHER OUTCOMES:
Anti-Mullerian Hormone levels variation | One year postoperatively
  Anti-Mullerian Hormone levels before surgery, 6 months and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Neset Gümüsburun, MD, Principal Investigator — Ataturk University
Locations (1):
- Atatürk Üniversitesi Araştırma Hastanesi, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Gumusburun N, Yapca OE, Ozdes S, Al RA. Triple vs. single uterine tourniquet to reduce hemorrhage at myomectomy: a randomized trial. Arch Gynecol Obstet. 2023 Dec;308(6):1811-1816. doi: 10.1007/s00404-023-07201-7. Epub 2023 Sep 6. PMID 37672088